CLINICAL TRIAL: NCT01901120
Title: Long-Term Specified Drug Use-results Survey of Betanis Tablets
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: BE0002
Record Dates: First submitted 2013-07-10; First posted 2013-07-17 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Overactive Bladder
Keywords: Betanis®; mirabegron; Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Betanis: the usual adult dosage of mirabegron once daily after a meal
  Interventions: Drug: Betanis

INTERVENTIONS:
Drug: Betanis — oral
  Other Names: YM178; mirabegron

SUMMARY:
This study is to evaluate the safety and efficacy of long-term use of Betanis (generic name: mirabegron), and to determine the adherence to treatment with mirabegron.

ELIGIBILITY:
Inclusion Criteria:

* Patients who administer mirabegron for treatment of urinary urgency, daytime frequency, and urgency incontinence associated with overactive bladder and also who have no treatment history of mirabegron.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who administer mirabegron for treatment of urinary urgency, daytime frequency, and urgency incontinence associated with overactive bladder and also who have no treatment history of mirabegron.
Sampling Method: Non-Probability Sample
Enrollment: 1263 (Actual)
Dates: Start 2012-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | Up to 36 months after treatment

SECONDARY OUTCOMES:
Overactive Bladder Symptom Score (OABSS) | At the start of treatment and 3, 6, 12, 18, 24, 30, and 36 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chūbu, Chubu
  - Chugoku, Chugoku
  - Hokkaido, Hokkaido
  - Kansai, Kansai
  - Kanto, Kanto
  - Kyushu, Kyushu
  - Shikoku, Shikoku
  - Tōhoku, Tohoku